CLINICAL TRIAL: NCT03498859
Title: Efficacy of Physiotherapist-supervised Rehabilitation After Two-part Proximal Humerus Fractures Treated Non-operatively. A Randomised Controlled Trial
Brief Title: Efficacy of Physiotherapist-supervised Rehabilitation After Proximal Humerus Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Tampere University Hospital (Other); Oslo University Hospital (Other); Regionshospitalet Viborg, Skive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProxHumRehab
Record Dates: First submitted 2018-04-03; First posted 2018-04-17 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Proximal Humeral Fracture
Keywords: Rehabilitation
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based training (Other): 10 weeks of home-based training with no supervision of a physiotherapist
  Interventions: Other: Home-based training
- Physiotherapist-supervised training (Other): Physiotherapist-supervised training once per week during 10 weeks in addition to home-based training
  Interventions: Other: Physiotherapist-supervised training

INTERVENTIONS:
Other: Physiotherapist-supervised training — The intervention is physiotherapist-supervised training once per week during 10 weeks.
  Arms: Physiotherapist-supervised training
Other: Home-based training — The intervention is home-based training during 10 weeks
  Arms: Home-based training

SUMMARY:
This study investigates the efficacy of physiotherapist-supervised training once per week during 10 weeks compared to home-based training during 10 weeks, after proksimal humerus fracture.

DETAILED DESCRIPTION:
Proximal humerus fracture is the third most common fracture in elderly people after hip and colles fracture, and are often caused by fall and osteoporosis. These fractures are highly related to morbidity and mortality among elderly people and consumes considerably health care resources. More than 70% of the proximal humerus fracture patients are over 60 years of age and 75% are female.

Only sparse evidence reveals to what extend the patients need rehabilitation and how it should be implemented in the treatment strategy.

In Denmark as well as in Finland the rehabilitation after proximal humerus fractures takes place in local centers in the municipalities, and the rehabilitation offered to the patients varies significantly. Currently in Denmark there are no national clinical guidelines to support the rehabilitation strategy.

ELIGIBILITY:
Inclusion Criteria:

•Low energy proximal humeral displaced (more than 5mm or 30 degrees) two-part fracture where fracture line emerges through the surgical (or anatomical) neck, treated non-operatively

Exclusion Criteria:

* Refuse to participate in the study
* Younger than 60 years old
* Non-independent
* Demented
* Does no understand written and spoken guidance in local language
* Pathological fracture or previous fracture in the same proximal humerus
* Other operational injuries in the same upper limb
* Major nerve injury (e.g. Complete radialis- or delta palsy)
* Open fracture
* Multi-trauma patient
* Fracture dislocation or head splitting fracture
* Undisplaced fracture
* Isolated tuberculum fracture
* Fracture has no precondition to ossify by conservative treatment (no bony contact between fracture parts or the humeral shaft is in contact with the articular surface)
* Treating surgeon considers patient unsuitable to attend the study on medical basis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
The Disability of the Arm, Shoulder and Hand (DASH) | Measured at 3 months after fracture
  Patient reported outcome measure of physical function in the upper extremity. Measures on a 0-100 scale, where a higher score indicates greater disability.
  The scores will be compared between the 2 groups

SECONDARY OUTCOMES:
The Disability of the Arm, Shoulder and Hand (DASH) | Measured at baseline and after 12 months
  Patient reported outcome measure of physical function in the upper extremity. Measures on a 0-100 scale, where a higher score indicates greater disability.
  The scores will be compared between the 2 groups
Constant Murley Shoulder Score | Measured after 3 and 12 months.
  Subjective and objective measurement of the shoulder function. Measures on a 0-100 scale, where a lower score indicates greater disability. The scores will be compared between the 2 groups
15-dimentional health-realted quality of life instrument (15D) | Measured at baseline, after 3 and 12 months
  Patient reported outcome measure of health related quality of life. A set of utility or preference weights is used to generate the 15D score (single index number) on a 0-1 scale, where a higher score indicates a poor health related quality of life.
  The scores will be compared between the 2 groups
Pain catastrophizing Scale | Measured at baseline, after 3 and 12 months
  Patient reported outcome measure. Measures on a 0-53 scale, where a higher score indicates a higher levels of pain catastrophizing thinking.
  The scores will be compared between the 2 groups. Also the correlation with DASH scores will be investigated
Generel Self-Efficacy scale | Measured at baseline, after 3 and 12 months
  Patient reported outcome measure. Measures on a 10-40 scale, where a higher score indicates a higher degree of self-efficacy.
  The scores will be compared between the 2 groups. Also the correlation with DASH scores will be investigated
Accelerometer based activity in the upper extremity | Measured at 3 and 12 months
  The patient is wearing a censor above the elbow on both arms, that measures the level of upper extremity activity for three consecutive days. It measures the number of movements under and above shoulder hight and classify them into either high or low intensity movements.
  The asymmetry between the fractured and the healthy arm will be estimated and compared between the groups.

OTHER OUTCOMES:
Follow up of the decliners | Measured at baseline and 3 months
  Patients declining to participate in the randomised trial will be invited to follow up visits, consisting of x-rays and identical questionnaires as used in the RCT
Cost-effectiveness | After 12 months
  A cost-effectiveness analysis (QALY) of the two training modalities will be performed and a ratio will be estimated.

CONTACTS AND LOCATIONS:
Locations (2):
- Viborg Regional Hospital, Viborg, Denmark
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196